CLINICAL TRIAL: NCT03665272
Title: Evaluation of the Effects of Different Fixation Methods on Wound Healing After Deepithelialized Gingival Graft
Brief Title: The Evaluation of the Deepithelialized Gingival Graft Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Zekeriya Tasdemir, Pricipal investigator, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Zeck
Record Dates: First submitted 2018-09-05; First posted 2018-09-11 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Wound Heal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fixation by tissue adhesive (Experimental): In this group, deepithelialized gingival grafts were fixed by tissue adhesive without any suture.
  Interventions: Procedure: deepithelialized gingival graft fixation
- fixation by sutures (Experimental): In this groups, deepithelialized gingival grafts were fixed by 4.0 round vicryl sutures.
  Interventions: Procedure: deepithelialized gingival graft fixation

INTERVENTIONS:
Procedure: deepithelialized gingival graft fixation — one group's deepithelialized gingival graft fixed by sutures and other one's by tissue adhesive.

SUMMARY:
The aim of this study was to compare of the effects of different fixation methods on deepithelialized gingival graft wound healing. Laser doppler flowmetry method was used to determine for blood perfusion changes. 40 patients were devided into two groups randomly and deepithelialized gingival graft procedure was performed and healings were evaluated by laser doppler flowmetry.

DETAILED DESCRIPTION:
This study evaluates the effects of different fixation methods on the early healing period of deepithelialized gingival grafts placed for non-root coverage gingival augmentation by laser Doppler flowmetry Forty patients were assigned to study groups: 1)test : tissue adhesive or 2) control group: suture. Forty patients completed the study. Blood perfusion in the recipient site was measured by laser doppler flowmetry on the day of surgery and at 3 and 7 days after surgery. Quality of life and pain at recipient sites were also investigated.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age
* systemically healthy
* inadequate amount or absence of keratinized gingiva on the labial side of the lower incisor region
* no restorations on the lower incisor region
* no mucogingival surgical history in the lower incisor region
* no periodontal treatment within the previous year
* no systemic antibiotics taken for 6 months before the study
* not pregnant or lactating
* no-smoking

Exclusion Criteria:

* lower 18 and upper than 65 years of age
* systemical disease
* adequate amount of keratinized gingiva on the labial side of the lower incisor region
* restorations on the lower incisor region
* mucogingival surgical history in the lower incisor region
* periodontal treatment within the previous year
* systemic antibiotics taken for ‡6months before the study
* pregnancy or lactating
* smoking history or current smokers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-09-03 (Actual); Study Completion 2018-09-03 (Actual)

PRIMARY OUTCOMES:
deepithelialized gingival graft blood perfusion change | measurements were performed at the day of surgery, 1, 3 and 7 days.
  Blood perfusions (units) were measured by laser doppler flowmetry

SECONDARY OUTCOMES:
Deepithelialized gingival graft recipient bed pain changes | measurements were performed at 1, 3 and 7 days post surgery.
  In this evaluations, we did not evaluate the total range we used subscale pain evaluation by visual analog scale. visual analog scale consisted of 10 units,in combination with a graphic rating scale.On the visual analog scale,the left and right end of the graphic represented the absence of pain (minimum 0)(score 0) and the most severe pain (maximum 10) (score 10),respectively. Patients were warned to complete the visual analog scale taking into consideration the intensity of their pain in the previous 24 hours on all recall days

CONTACTS AND LOCATIONS:
Overall Officials: zekeriya taşdemir, phd, Principal Investigator — TC Erciyes University
Locations (1):
- Zekeriya Taşdemir, Kayseri, Melikgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided